CLINICAL TRIAL: NCT00185588
Title: A Phase 1-2 Study of the VEGF Receptor Tyrosine Kinase Inhibitor PTK787/ZK 222584 <Vatalanib> and Gemcitabine in Patients With Advanced Pancreatic Cancer
Brief Title: Phase 1-2 Vatalanib and Gemcitabine in Advanced Pancreatic Cancer
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: George Albert Fisher (Other)
Collaborators: Novartis (Industry)
Responsible Party: Sponsor-Investigator, George Albert Fisher, Associate Professor of Medicine, Stanford University
Organization: Stanford University (Other)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IRB-06999; 95533 (Other: Stanford University Alternate IRB Number); CPTK787AUS08 (Other: Novartis); PANC0002 (Other: OnCore)
Record Dates: First submitted 2005-09-12; First posted 2005-09-16 (Estimated); Results first posted 2014-09-15 (Estimated); Last update posted 2014-09-15 (Estimated); Status verified 2014-09

CONDITIONS: Pancreatic Cancer
MeSH Terms: conditions — Pancreatic Neoplasms | interventions — vatalanib; Gemcitabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Stage 1 Dose Exploration 0 - Gemcitabine 700 + vatalanib 1250 (Experimental): Gemcitabine 700 mg/m2 + vatalanib 1250 mg daily
  Interventions: Drug: Vatalanib; Drug: Gemcitabine
- Stage 1 Dose Exploration 1 - Gemcitabine 850 + vatalanib 1250 (Experimental): Gemcitabine 850 mg/m2 + vatalanib 1250 mg
  Interventions: Drug: Vatalanib; Drug: Gemcitabine
- Stage 1 Dose Explrtion2 - Gemcitabine850+vatalanib 2x250/2x500 (Experimental): Gemcitabine 850 mg/m2 + vatalanib 250 mg Q12 hours x 1 week then 500 mg Q12 hours thereafter
  Interventions: Drug: Vatalanib; Drug: Gemcitabine
- Stage 2 Dose Expansion - Gemcitabine850+vatalanib 2x250/2x500 (Experimental): Gemcitabine 850 mg/m2 + vatalanib 250 mg Q12 hours x 1 week then 500 mg Q12 hours thereafter
  Interventions: Drug: Vatalanib; Drug: Gemcitabine

INTERVENTIONS:
Drug: Vatalanib — Vatalanib 250 mg PO Q12 hours x 7 days, 8th day forward 500 mg PO Q12 hours
  Other Names: PTK787; ZK 222584; PTK787/ZK 222584
Drug: Gemcitabine — 850 mg/m2
  Other Names: Gemzar

SUMMARY:
The purpose of the study is to determine the optimal safe and tolerable dose of gemcitabine in combination with once daily or twice daily dose of PTK/ZK in patients with unresectable pancreatic cancer. The Phase II part of this study planned to determine the antitumor activity of this regimen and its effectiveness of preventing tumor growth and spread.

ELIGIBILITY:
Inclusion Criteria

* Histologically or cytologically confirmed adenocarcinoma of the pancreas
* Unresectable (due to involvement of critical vasculature, adjacent organ invasion, or presence of metastasis)
* If > 5 years between the primary surgery and the development of metastatic disease, then separate histological or cytological confirmation of metastatic disease
* Primary or metastatic lesion within 4 weeks prior to entry of study
* WHO performance status of 0 to 2
* ≤ 18 years of age
* Absolute Neutrophil Count (ANC) ≥ 1.5 x 10e9/L (>= 1500/mm3)
* Platelets (PLT) ≥ 100 x 10^9/L (≥ 100,000/mm3)
* Hemoglobin (Hgb) ≥ 9 g/dL
* Serum creatinine ≤ 1.5 upper limit of normal (ULN)
* Serum bilirubin ≤ 1.5 ULN
* Aspartate aminotransferase (AST/SGOT) and alanine aminotransferase

  * (ALT/SGPT) ≤ 3.0 x ULN OR
  * ≤ 5 x ULN if liver metastases present
* Proteinuria:

  * Negative for proteinuria based on dip stick reading OR
  * If dip stick reading is +1 result, then total urinary protein ≤ 500 mg and measured creatinine clearance (CrCl) ≥ 50 mL/min from a 24-hour urine collection
* Life expectancy ≥ 12 weeks
* Ability to give written informed consent

Exclusion Criteria

* For the "phase 1" portion of the study: prior gemcitabine will be therapy.
* For the "phase 2" portion of the study: any prior chemotherapy {except for low-dose 5-fluorouracil (5-FU)as a radiosensitizer]
* Radiotherapy (RT). The site of previous RT must have progressive disease if the only site of disease).

  * Prior full field radiotherapy ≤ 4 weeks prior to enrollment OR
  * Limited field radiotherapy ≤ 2 weeks prior to enrollment. Patients must have recovered from all therapy-related toxicities.
* Prior biologic or immunotherapy ≤ 2 weeks prior to registration.
* Prior therapy with anti-VEGF agents
* History or presence of central nervous system (CNS) disease
* Patients with a history of another primary malignancy ≤ 5 years (Exception: inactive basal or squamous cell carcinoma of the skin)
* Major surgery ≤ 4 weeks prior to enrollment. (Exception: insertion of a vascular access device)
* Minor surgery ≤ 2 weeks prior to enrollment. (Exception: insertion of a vascular access device)
* Concurrent use of other investigational agents and patients who have received investigational drugs ≤ 4 weeks prior to enrollment.
* Pregnant, or breast-feeding, not employing an effective method of birth control.
* Pre-existing peripheral sensory neuropathy with functional impairment (≥ CTCAE grade 2 neuropathy)
* Respiratory compromise due to pleural effusion or ascites (≥ CTCAE grade 2 dyspnea)
* QTc > 450 ms (male) or > 470 ms (female)
* Uncontrolled high blood pressure
* History of labile hypertension
* History of poor compliance with an antihypertensive regimen
* Unstable angina pectoris
* Symptomatic congestive heart failure
* Myocardial infarction ≤ 6 months prior to registration / randomization
* Serious uncontrolled cardiac arrhythmia
* Uncontrolled diabetes
* Active or uncontrolled infection
* Interstitial pneumonia
* Extensive and symptomatic interstitial fibrosis of the lung
* Chronic renal disease
* Acute or chronic liver disease
* Impairment of gastrointestinal (GI) function or GI disease that may significantly alter the absorption of vatalanib
* Human immunodeficiency virus (HIV) infection (confirmed), if there is potential for interaction between vatalanib and any anti-HIV medication
* HIV infection (confirmed) judged to increase subject risk due to the pharmacologic activity of vatalanib
* Receiving warfarin sodium (Coumadin) or similar. Heparin is allowed.
* Unwilling to or unable to comply with

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 33 (Actual)
Dates: Start 2004-10; Primary Completion 2009-01 (Actual); Study Completion 2009-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: George Albert Fisher M.D. Ph.D., Principal Investigator — Stanford University
Locations (1):
- Stanford University School of Medicine, Stanford, California, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Stage 1 Dose Exploration 0 - Gemcitabine 700 + Vatalanib 1250: Gemcitabine 700 mg/m2 + vatalanib 1250 mg daily
  Vatalanib: Vatalanib 250 mg PO Q12 x 7 days, 8th day forward 500 mg PO Q12
  Gemcitabine: 850 mg/m2
- Stage 1 Dose Exploration 1 - Gemcitabine 850 + Vatalanib 1250: Gemcitabine 850 mg/m2 + vatalanib 1250 mg
  Vatalanib: Vatalanib 250 mg PO Q12 x 7 days, 8th day forward 500 mg PO Q12
  Gemcitabine: 850 mg/m2
- Stage 1 Dose Explrtion2 - Gemcitabine850+Vatalanib 2x250/2x500: Gemcitabine 850 mg/m2 + vatalanib 250 mg Q12 hours x 1 week then 500 mg Q12 hours thereafter
  Vatalanib: Vatalanib 250 mg PO Q12 x 7 days, 8th day forward 500 mg PO Q12
  Gemcitabine: 850 mg/m2
- Stage 2 Dose Expansion - Gemcitabine850+Vatalanib 2x250/2x500: Gemcitabine 850 mg/m2 + vatalanib 500 mg twice daily
  Vatalanib: Vatalanib 250 mg PO Q12 x 7 days, 8th day forward 500 mg PO Q12
  Gemcitabine: 850 mg/m2
Period: Overall Study
Arm/Group | Stage 1 Dose Exploration 0 - Gemcitabine 700 + Vatalanib 1250 | Stage 1 Dose Exploration 1 - Gemcitabine 850 + Vatalanib 1250 | Stage 1 Dose Explrtion2 - Gemcitabine850+Vatalanib 2x250/2x500 | Stage 2 Dose Expansion - Gemcitabine850+Vatalanib 2x250/2x500
Started | 6 | 4 | 6 | 17
Completed | 3 | 2 | 0 | 13
Not Completed | 3 | 2 | 6 | 4
Not completed — Adverse Event | 3 | 1 | 4 | 2
Not completed — Lost to Follow-up | 0 | 0 | 1 | 2
Not completed — Withdrawal by Subject | 0 | 1 | 0 | 0
Not completed — Physician Decision | 0 | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Population: 33 adult patients with advanced pancreatic cancer
Groups:
- Total: Total of all reporting groups
Arm/Group | Stage 1 Dose Exploration 0 - Gemcitabine 700 + Vatalanib 1250 | Stage 1 Dose Exploration 1 - Gemcitabine 850 + Vatalanib 1250 | Stage 1 Dose Explrtion2 - Gemcitabine850+Vatalanib 2x250/2x500 | Stage 2 Dose Expansion - Gemcitabine850+Vatalanib 2x250/2x500 | Total
Number analyzed (Participants) | 6 | 4 | 6 | 17 | 33
Age, Continuous [Median (Full Range); unit: years] | 55 [40 to 76] | 69 [53 to 82] | 70 [53 to 75] | 55 [40 to 79] | 58 [40 to 82]
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 5 | 2 | 2 | 13 | 22
  >=65 years | 1 | 2 | 4 | 4 | 11
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 2 | 2 | 7 | 15
  Male | 2 | 2 | 4 | 10 | 18
Region of Enrollment [Number; unit: participants]
  United States | 6 | 4 | 6 | 17 | 33

OUTCOME MEASURES:

1. Primary Outcome: Time-to-Treatment Failure (Intent-To-Treat Analysis)
Description: For the purposes of an Intent-to-Treat (ITT) analysis, Time-to-Treatment Failure (TTF) was defined as the time from treatment initiation to treatment discontinuation for any reason, including disease progression, treatment toxicity, patient preference, lost-to-follow-up, or death.
  Progression was defined using Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.0).
Time Frame: 12 months
Measure: Median (Full Range); unit: months
Arm/Group | Stage 1 Dose Exploration 0 - Gemcitabine 700 + Vatalanib 1250 | Stage 1 Dose Exploration 1 - Gemcitabine 850 + Vatalanib 1250 | Stage 1 Dose Explrtion2 - Gemcitabine850+Vatalanib 2x250/2x500 | Stage 2 Dose Expansion - Gemcitabine850+Vatalanib 2x250/2x500
Number analyzed (Participants) | 6 | 4 | 6 | 17
months | 4.9 [3.8 to 9.5] | 2.7 [0.7 to 9.8] | 2.2 [0.7 to 5.6] | 3.7 [0.7 to 10.4]

2. Secondary Outcome: Time-to-Progression, Evaluable Patients
Description: Represents the evaluable subset of subjects that terminated from the study due to disease progression (endpoint). Does not include any other form of treatment failure, nor lost-to-follow-up.
Time Frame: 12 months
Population: Evaluable subset of subjects that terminated from the study due to disease progression (endpoint).
  No participants were analyzed in the "Stage 1 Dose Exploration 2 - Gemcitabine 850 + Vatalanib 2 x 250 / 2 x 500 group" because no evaluable participants progressed within 12 months.
Measure: Median (Full Range); unit: months
Arm/Group | Stage 1 Dose Exploration 0 - Gemcitabine 700 + Vatalanib 1250 | Stage 1 Dose Exploration 1 - Gemcitabine 850 + Vatalanib 1250 | Stage 1 Dose Explrtion2 - Gemcitabine850+Vatalanib 2x250/2x500 | Stage 2 Dose Expansion - Gemcitabine850+Vatalanib 2x250/2x500
Number analyzed (Participants) | 3 | 2 | 0 | 13
months | 4.4 [3.8 to 6.0] | 6.0 [2.1 to 9.8] |  | 3.2 [0.7 to 8.3]

ADVERSE EVENTS:
Arm/Group | Stage 1 Dose Exploration 0 - Gemcitabine 700 + Vatalanib 1250 | Stage 1 Dose Exploration 1 - Gemcitabine 850 + Vatalanib 1250 | Stage 1 Dose Explrtion2 - Gemcitabine850+Vatalanib 2x250/2x500 | Stage 2 Dose Expansion - Gemcitabine850+Vatalanib 2x250/2x500
Serious Adverse Events (participants affected / at risk) | 6/6 | 4/4 | 4/6 | 10/17
Other Adverse Events (participants affected / at risk) | 6/6 | 3/4 | 6/6 | 14/17
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Stage 1 Dose Exploration 0 - Gemcitabine 700 + Vatalanib 1250 (N=6) | Stage 1 Dose Exploration 1 - Gemcitabine 850 + Vatalanib 1250 (N=4) | Stage 1 Dose Explrtion2 - Gemcitabine850+Vatalanib 2x250/2x500 (N=6) | Stage 2 Dose Expansion - Gemcitabine850+Vatalanib 2x250/2x500 (N=17)
Anemia (Blood and lymphatic system disorders) | 1 (1) | 1 (2) | 0 (0) | 1 (2)
Febrile neutropenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Hemolysis (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 4 (4)
Abdominal pain-intractable pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Ascites (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Colitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Constipation (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Diarrhea (Gastrointestinal disorders) | 2 (3) | 0 (0) | 0 (0) | 0 (0)
Dyspepsia (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Enterocolitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Gastritis (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hemorrhoids (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Rectal hemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Vomiting (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Edema limbs (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Fatigue (General disorders) | 2 (3) | 0 (0) | 1 (1) | 0 (0)
Fever (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Obstructed bile duct, stent placement (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Neutropenia ANC 210 (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Bladder (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Infections and infestations - not specified (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Urinary tract NOS (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Urosepsis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Lung Infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Urinary tract infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Arterial injury (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Vascular access complication (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Alanine aminotransferase increased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Alkaline phosphatase increased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Blood bilirubin increased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Neutrophil count decreased (Investigations) | 2 (4) | 1 (1) | 1 (1) | 2 (3)
Platelet count decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
White blood cell decreased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Anorexia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 2 (2) | 0 (0) | 0 (0) | 1 (1)
Hyperglycemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hypokalemia (Metabolism and nutrition disorders) | 2 (3) | 0 (0) | 0 (0) | 0 (0)
Hyponatremia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Peripheral sensory neuropathy (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Proteinuria (Renal and urinary disorders) | 1 (2) | 0 (0) | 1 (2) | 0 (0)
Urinary tract obstruction (Renal and urinary disorders) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hypertension (Vascular disorders) | 1 (1) | 1 (2) | 0 (0) | 0 (0)
Thromboembolic event (Vascular disorders) | 2 (2) | 0 (0) | 1 (1) | 0 (0)
Thromboembolic event-DVT (Vascular disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Stage 1 Dose Exploration 0 - Gemcitabine 700 + Vatalanib 1250 (N=6) | Stage 1 Dose Exploration 1 - Gemcitabine 850 + Vatalanib 1250 (N=4) | Stage 1 Dose Explrtion2 - Gemcitabine850+Vatalanib 2x250/2x500 (N=6) | Stage 2 Dose Expansion - Gemcitabine850+Vatalanib 2x250/2x500 (N=17)
Anemia (Blood and lymphatic system disorders) | 4 (13) | 1 (4) | 3 (3) | 5 (12)
Febrile neutropenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1) | 2 (2)
Cardiac disorders - not specified (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Ear and labyrinth disorders-not specified (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Blurred vision (Eye disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Abdominal distension (Gastrointestinal disorders) | 1 (1) | 1 (1) | 3 (3) | 1 (7)
Abdominal pain (Gastrointestinal disorders) | 6 (11) | 0 (0) | 1 (1) | 10 (16)
Constipation (Gastrointestinal disorders) | 4 (6) | 0 (0) | 1 (1) | 9 (10)
Diarrhea (Gastrointestinal disorders) | 3 (6) | 0 (0) | 1 (1) | 3 (6)
Dyspepsia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 2 (2) | 3 (6)
Esophagitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Flatulence (Gastrointestinal disorders) | 1 (2) | 0 (0) | 0 (0) | 1 (1)
Gastric stenosis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Gastric ulcer (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Gastritis (Gastrointestinal disorders) | 1 (2) | 1 (1) | 1 (1) | 1 (1)
Gastrointestinal disorders -not specified (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 3 (3)
Hemorrhoids (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Mucositis oral (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Nausea (Gastrointestinal disorders) | 3 (4) | 1 (1) | 2 (2) | 12 (17)
Stomach pain (Gastrointestinal disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Toothache (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Vomiting (Gastrointestinal disorders) | 2 (2) | 0 (0) | 1 (2) | 6 (9)
Chills (General disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (3)
Edema face (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Edema limbs (General disorders) | 1 (1) | 0 (0) | 1 (1) | 1 (1)
Fatigue (General disorders) | 3 (6) | 2 (4) | 4 (7) | 11 (17)
Fever (General disorders) | 4 (5) | 0 (0) | 1 (2) | 3 (6)
Injection site reaction (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pain (General disorders) | 1 (1) | 0 (0) | 0 (0) | 2 (6)
Hepatic failure (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Urinary tract NOS (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 2 (2)
Skin infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Bruising (Injury, poisoning and procedural complications) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Vascular access complication (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Wound dehiscence (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Alanine aminotransferase increased (Investigations) | 1 (6) | 0 (0) | 2 (2) | 3 (5)
Alkaline phosphatase increased (Investigations) | 1 (1) | 1 (1) | 1 (2) | 5 (7)
Aspartate aminotransferase increased (Investigations) | 1 (1) | 0 (0) | 2 (2) | 6 (10)
Blood bilirubin increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Creatinine increased (Investigations) | 0 (0) | 0 (0) | 2 (3) | 0 (0)
INR increased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Neutrophil count decreased (Investigations) | 5 (11) | 3 (6) | 2 (3) | 5 (6)
Platelet count decreased (Investigations) | 4 (9) | 1 (3) | 3 (3) | 5 (9)
Weight gain (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Weight loss (Investigations) | 0 (0) | 0 (0) | 0 (0) | 3 (3)
White blood cell decreased (Investigations) | 3 (13) | 0 (0) | 2 (2) | 5 (6)
Anorexia (Metabolism and nutrition disorders) | 4 (5) | 0 (0) | 2 (2) | 6 (7)
Dehydration (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 2 (2)
Hyperglycemia (Metabolism and nutrition disorders) | 1 (7) | 0 (0) | 1 (1) | 0 (0)
Hyperkalemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hypoalbuminemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (2) | 3 (4)
Hypoglycemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hypokalemia (Metabolism and nutrition disorders) | 1 (3) | 0 (0) | 1 (1) | 0 (0)
Hyponatremia (Metabolism and nutrition disorders) | 1 (3) | 0 (0) | 0 (0) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 4 (4) | 0 (0) | 1 (1) | 5 (5)
Chest wall pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 1 (1) | 1 (1)
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Muscle weakness lower limb (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Musculoskeletal and connective tissue disorder-not specified (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Neck pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 3 (3) | 0 (0) | 3 (3) | 0 (0)
Trismus (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Dizziness (Nervous system disorders) | 1 (1) | 0 (0) | 1 (1) | 2 (3)
Headache (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 2 (2)
Memory impairment (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Nervous system disorders - not specified (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Peripheral motor neuropathy (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Syncope (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Tremor (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Anxiety (Psychiatric disorders) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
Confusion (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Depression (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 3 (3)
Insomnia (Psychiatric disorders) | 0 (0) | 1 (1) | 2 (3) | 3 (3)
Cystitis noninfective (Renal and urinary disorders) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
Proteinuria (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) | 2 (2)
Renal and urinary disorders - not specified (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Urine discoloration (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Pelvic pain (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) | 3 (5) | 1 (1)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0) | 2 (2) | 4 (4)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 2 (2)
Hiccups (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Pleuritic pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Sinus disorder (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0) | 0 (0) | 1 (1)
Voice alteration (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Alopecia (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 2 (2) | 0 (0) | 1 (2) | 0 (0)
Pain of skin (Skin and subcutaneous tissue disorders) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (3) | 0 (0) | 3 (5)
Skin and subcutaneous tissue disorders - not specified (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hypertension (Vascular disorders) | 0 (0) | 0 (0) | 1 (1) | 4 (5)
Hypotension (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Phlebitis (Vascular disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Thromboembolic event (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No